CLINICAL TRIAL: NCT05480709
Title: Evaluation Der Unmittelbaren Und Mittelfristigen Gesundheits- Und Arbeitsbezogenen Effekte in Folge Einer Stationären Psychokardiologischen Rehabilitation [Evaluation of Immediate and Medium-term Health- and Work-related Effects Following Inpatient Psychocardiological Rehabilitation]
Brief Title: Evaluation of Immediate and Medium-term Health- and Work-related Effects Following Inpatient Psychocardiological Rehabilitation
Acronym: EvalPsyKard
Status: Completed | Type: Observational
Sponsor: Pensionsversicherungsanstalt (Other)
Responsible Party: Sponsor
Other Study IDs: 0005 Evaluation PsyKard
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Psychiatric Disorder
Keywords: Psychocardiology; Rehabilitation; Observational Study; Return to Work
MeSH Terms: conditions — Cardiovascular Diseases; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Psychocardiological Rehabilitation — Psychocardiological Rehabilitation: Regular cardiac rehabilitation with in-depth psychological and psychotherapeutic care, individual and group counseling, relaxation training, and interdisciplinary specialist psychiatric and psychosomatic visits.

SUMMARY:
Since May 2019, psychocardiological rehabilitation has been carried out at the Rehabilitation Center Felbring (RFE) in the form of a pilot project. The background is the mutual relationship of psychological and physical morbidity, which is of particular importance in cardiological rehabilitation. The present outcome evaluation study is designed as a quantitative longitudinal study with 4 repeated measures, in which at least 75 rehabilitation patients will be included. Three assessments are conducted at admission and discharge to/from inpatient rehabilitation, and an additional survey will be conducted by mail 6 months after the end of rehabilitation. Effects that become apparent as a result of rehabilitation will be recorded from a patient-centered perspective by means of "patient-reported outcomes". In this way, primarily psychological and work-related changes, but also changes in the physical quality of life are to be mapped, which can be determined immediately after completion of rehabilitation and continue in the medium term up to 6 months later.

ELIGIBILITY:
Inclusion Criteria:

Cardiovascular disease and increased psychological distress due to one of the following mental health diagnoses (according to ICD-10):

* Depressive Episode
* Recurrent depressive disorder
* Phobic disorders
* Anxiety disorders (incl. panic disorder)
* Acute stress reaction
* Post-traumatic stress disorder
* Adjustment disorders
* Other reactions to severe stress
* Psychological or behavioral factors that play a significant role in the etiology of physical illnesses

Exclusion Criteria:

* Acute danger to self or others
* Acute mental disorders, the extent and/or instability of which does not allow participation in rehabilitation
* High degree of neurocognitive deficits
* Highly degraded communication skills

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — "male", "female", "diverse"
Study Population: Employed rehabilitation patients with cardiological and psychiatric illness in inpatient rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Symptom-Checklist-90 - Standard (SCL-90-S) | 6 weeks of inpatient rehabilitation with follow-up assessment 6 months after rehabilitation.
  Psychological problems and symptoms of psychopathology. Minimum value (Global Severity Index) = 0. Maximum value (Global Severity Index) = 360. Lower values indicate better outcomes (i.e. less symptoms of psychopathology).
Herzangstfragebogen (HAF-17) | 6 weeks of inpatient rehabilitation with follow-up assessment 6 months after rehabilitation.
  [Cardiac Anxiety Questionnaire - German version] Heart-focused anxiety. Minimum value = 0. Maximum value = 4. Lower values indicate less heart-focused anxiety.
Short Form-12 Health Survey (SF-12) | 6 weeks of inpatient rehabilitation with follow-up assessment 6 months after rehabilitation.
  Health-related quality of life. Norm-based values (M = 50, SD = 10) for the Physical component scale (PCS) and Mental component scale (MCS). Values below 50 indicate below average (i.e. worse) physical or mental health-related quality of life. Values above 50 indicate above average (i.e. better) physical or mental health-related quality of life.
Subjective work ability | 6 weeks of inpatient rehabilitation with follow-up assessment 6 months after rehabilitation.
  Question "To what extent are you impaired in your work by your current state of health?", rated on a 10 point Likert scale, ranging from 0 = no impairment to 10 = total impairment. Lower values indicate better subjective work ability.
Employment status | 6 weeks of inpatient rehabilitation with follow-up assessment 6 months after rehabilitation.
  Nominal scale (Full-time employed, Employed at least part-time, Unemployed, Retired)

SECONDARY OUTCOMES:
Arbeitsbezogenes Verhaltens- und Erlebensmuster (AVEM) | 6 weeks of inpatient rehabilitation.
  [Work-related behavior and experience patterns (AVEM) - German version] Work-related behavioral health risks, resources and coping. Patients are classified into four work-related behavioral and experiential patterns: G (healthy pattern), S (unambitious pattern), A (pattern at risk for overexertion) and B (pattern at risk for chronic exhaustion and resignation). Pattern G (healthy pattern) is the desirable outcome.
Social Adjustment Scale Self-Report (SAS-SR) | 6 weeks of inpatient rehabilitation.
  Social adjustment / instrumental and expressive role performance at work, in social activities, and with family. Up to 54 items are rated on a five-point scale (1-5), summed and diveded by the number of items actually scored to obtain an overall mean. Lower scores indicate better social adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Stöhr, Mag., Study Chair — Pensionsversicherungsanstalt
Locations (1):
- Rehabilitationszentrum Felbring, Muthmannsdorf, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: No